CLINICAL TRIAL: NCT00295477
Title: A Phase I/II, Open-label, Single Center Study to Evaluate the Tolerability, Trafficking and Therapeutic Effects of Repeated Doses of Autologous T Cells Transduced With VRX496 in HIV Infected Subjects
Brief Title: Evaluate the Tolerability and Therapeutic Effects of Repeated Doses of Autologous T Cells With VRX496 in HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tebas 066290 - Protocol 802456; NIAID U19-A1066290 (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: HIV
Keywords: HIV; Treatment Experienced
MeSH Terms: interventions — lexgenleucel-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

INTERVENTIONS:
Genetic: VRX496 — In Step 1 of the protocol, each subject will receive up to 2 cycles of VRX496. Each treatment cycle consists of 3 infusions of VRX496.

SUMMARY:
The study is intended for individuals who are doing well on HAART therapy. In Step 1 of the trial, individuals will be given up to 6 infusions of the study drug VRX496 to see the effect on viral load and CD4 counts. If individuals have no serious adverse effects from the infusions of VRX496 and the viral load and CD4 counts remain stable, they may go on to Step 2 of the study. In Step 2, individuals will stop taking their HAART medication and their viral load, CD4 counts and the number of VRX496 in T cells will be monitored.

All subjects who receive VRX496 T cells will enroll in a Long-Term Follow-up study to monitor subjects. Subjects will be followed every 6 months for five years following the 1st infusion of the T cells. If the VRX496 T cells are no longer found in the blood after five years, then subjects will be contacted yearly for the next 10 years. If the VRX496 T cells are found in the blood at five years after the 1st infusion of T cells, then the subjects will continue to be seen once a year until the VRX496 T cells are no longer found in the blood for a maximum of 15 years.

DETAILED DESCRIPTION:
HIV-based antisense vectors may provide several important advantages over current HIV combination therapies. VIRxSYS Corporation (VIRxSYS) is developing the candidate clinical vector VRX496. VRX496 is an HIV-based lentiviral vector containing an anti-HIV antisense sequence targeted to the HIV envelope (env) coding sequence. First, HIV-1 vectors are likely to be less toxic than current combination drug therapies because the genetic antisense antiviral is expressed only in cells that become infected with wt-HIV. The payload is located upstream of a major splice acceptor site and is thus dependent on the expression of Tat and Rev proteins that are provided by wt-HIV. Second, the length of the antisense region is over 900 nucleotides long, making it difficult for wt-HIV to create resistant strains that are sufficiently fit to cause disease. Third, HIV vectors are predicted to be safe because no novel genetic sequences are introduced into the patient (i.e., no novel functional genes are contained in the HIV-1 vector). All the sequences present in the vector are derived from highly conserved regions of wt-HIV that would almost certainly be present in any HIV-1-infected individual. The HIV sequences that are used to create VRX496 are solely derived from pNL4-3, a prototypic HIV-1 molecular clone that is derived from two North American strains of HIV-1.

In the present trial, T cells will be harvested from infected individuals, transduced ex vivo with the vector at the University of Pennsylvania, and then reintroduced by autologous transfusions. VIRxSYS recently completed a Phase 1 clinical study at the University of Pennsylvania of the vector VRX496 in 5 HIV-positive subjects who had failed at least two HAART regimens. Data available to date for the primary endpoints, viral load and CD4 counts, are promising. Specifically, 4 of 5 subjects had stable or increased CD4 counts, and viral loads were stable in 4 of 5 patients, and decreased by 1.7 log in 1 of 5 subjects following a single infusion of VRX496 T cells. In the present trial, subjects will receive up to 6 infusions of VRX496 modified CD4 T cells, and then undergo a series of tests, including rectal mucosal biopsies, to determine the longevity and trafficking of the VRX496 T cells. In addition, subjects will have the opportunity to have a supervised drug holiday (structured treatment interruption) to determine if the VRX496 have an antiviral effect.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive by western blot or detection of HIV RNA in blood and responding to combination antiviral therapy
* No changes in antiretroviral medications within past 4 weeks of study entry and willing to continue on current therapy for the duration of the study
* 18 years of age and older
* Karnofsky Performance score of greater than 80
* HIV viral load < 59 copies/mL
* CD4 T cell count > 350 cells per uL
* adequate venous access

Exclusion Criteria:

* HIV seroconversion within past year
* History of cancer (other than a removed basal or squamous cell of the skin)
* History of congestive heart failure.
* Previous treatment with HIV experimental vaccine within past year
* Previous treatment with any gene therapy
* Positive serology for Vesicular Stomatitis Virus (VSV-G or VSV-G DNA)
* Currently breastfeeding, pregnant, or unwilling to use birth control
* Using oral corticosteroids, hydroxyurea, or immunomodulating agents (IL-2, interferon-gamma, granulocyte colony stimulating factors, megestrol acetate) within the past 30 days or foresee the need to use these during the study period.
* Are presently drug or alcohol dependent
* Have other serious illness or acute opportunistic infection or bacterial infection requiring systemic treatment and/or hospitalization within the past 30 days
* Have chronic hepatitis B or hepatitis C
* Have an active AIDS defining illness
* Have an allergy or hypersensitivity to human serum albumin, DMSO or Dextran 40
* Have diabetes or a coagulopathy with in the opinion of the investigator would exclude subjects from participating in rectal biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events & dose related toxicity. | 18 months
Effects on viral load and CD4 counts from baseline through STI. | 18 months
Estimate antiviral effects of VRX496 after STI. | 18 months

SECONDARY OUTCOMES:
Determine persistence and number of VRX496 containing T cells | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Tebas P, Stein D, Binder-Scholl G, Mukherjee R, Brady T, Rebello T, Humeau L, Kalos M, Papasavvas E, Montaner LJ, Schullery D, Shaheen F, Brennan AL, Zheng Z, Cotte J, Slepushkin V, Veloso E, Mackley A, Hwang WT, Aberra F, Zhan J, Boyer J, Collman RG, Bushman FD, Levine BL, June CH. Antiviral effects of autologous CD4 T cells genetically modified with a conditionally replicating lentiviral vector expressing long antisense to HIV. Blood. 2013 Feb 28;121(9):1524-33. doi: 10.1182/blood-2012-07-447250. Epub 2012 Dec 20. PMID 23264589
- See also: Click here for more information about this study under Clinical Trials — http://www.uphs.upenn.edu/pennactu/